CLINICAL TRIAL: NCT05519878
Title: Assessing Efficacy of a Light Therapy and Occupational Therapy Fatigue Management-Based Intervention for Patients With Genitourinary Cancers
Brief Title: Light Therapy and Occupational Therapy Fatigue Management-Based Intervention for Patients With Genitourinary Cancers
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: City of Hope Medical Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Factorial | Masking: None | Purpose: Supportive Care
Other Study IDs: 22235; NCI-2022-05658 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 22235 (Other: City of Hope Medical Center); P30CA033572 (NIH)
Record Dates: First submitted 2022-08-22; First posted 2022-08-29 (Actual); Last update posted 2025-12-24 (Actual); Status verified 2025-12

CONDITIONS: Bladder Carcinoma; Genitourinary System Neoplasm; Kidney Carcinoma; Prostate Carcinoma
MeSH Terms: conditions — Urinary Bladder Neoplasms; Carcinoma, Renal Cell; Prostatic Neoplasms | interventions — Practice Guidelines as Topic; Standard of Care; Ultraviolet Therapy; Occupational Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (4):
- Arm I (BWL) (Experimental): Patients self-administer 30 minutes of light delivered via light glasses every morning for 3 months. Patients attend 6 follow up sessions to address any questions regarding the wearable light therapy glasses.
  Interventions: Device: Bright White Light Therapy; Other: Questionnaire Administration
- Arm II (OT) (Experimental): Patients undergo 6 occupational therapist-led sessions over 60 minutes each.
  Interventions: Behavioral: Occupational Therapy; Other: Questionnaire Administration
- Arm III (OT, BWL) (Experimental): Patients self-administer 30 minutes of light delivered via light glasses every morning for 3 months. Patients attend 6 follow up sessions to address any questions regarding the wearable light therapy glasses and to complete the occupational therapist-led session over 60 minutes.
  Interventions: Device: Bright White Light Therapy; Behavioral: Occupational Therapy; Other: Questionnaire Administration
- Arm IV (Control) (Active Comparator): Patients undergo routine treatment and usual follow up care with their medical oncologist.
  Interventions: Other: Best Practice; Other: Questionnaire Administration

INTERVENTIONS:
Other: Best Practice — Undergo routine treatment and usual follow up care
  Other Names: standard of care; standard therapy
  Arms: Arm IV (Control)
Device: Bright White Light Therapy — Undergo bright white therapy
  Other Names: Bright Light Therapy; Bright White Light; BWL
  Arms: Arm I (BWL); Arm III (OT, BWL)
Behavioral: Occupational Therapy — Undergo occupational therapy
  Other Names: OT
  Arms: Arm II (OT); Arm III (OT, BWL)
Other: Questionnaire Administration — Complete questionnaires

SUMMARY:
This clinical trial evaluates light therapy and occupational therapy in improving cancer related fatigue (CRF) patients with genitourinary cancers. Light therapy is a non-pharmacological and evidence-based intervention for managing fatigue in cancer patients. The use of light therapy can provide a low burden, inexpensive, and easy to disseminate intervention approach that can potentially have a larger impact on CRF. In addition, occupational therapy is a standard, but often underutilized, component of the multi-disciplinary approach to cancer care. Using the combination of light therapy and occupational therapy may be effective in CRF management.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVE:

I. To evaluate patient's fatigue at post-intervention (3 months from baseline).

SECONDARY OBJECTIVE:

I. To evaluate whether the change (improvement) in fatigue as measured by the Functional Assessment of Chronic Illness Therapy (FACIT)-Fatigue tool, from pre-interventions to post interventions is significantly different between intervention groups in patients with genitourinary cancers.

THIRD OBJECTIVE:

I. To assess patient perceived changes in occupational performance as measured by the Canadian Occupational and Performance Measure (COPM) tool, in the occupational therapy (OT) group, compared to the control group in patients with genitourinary cancers.

OUTLINE: Patients are randomized to 1 of 4 arms.

ARM I (Bright white light [BWL]): Patients self-administer 30 minutes of light delivered via light glasses every morning for 3 months. Patients attend 6 follow up sessions to address any questions regarding the wearable light therapy glasses.

ARM II (OT): Patients undergo 6 occupational therapist-led sessions over 60 minutes each.

ARM III (BWL and OT): Patients self-administer 30 minutes of light delivered via light glasses every morning for 3 months. Patients attend 6 follow up sessions to address any questions regarding the wearable light therapy glasses and to complete the occupational therapist-led session over 60 minutes.

ARM IV (CONTROL): Patients undergo routine treatment and usual follow up care with their medical oncologist.

After completion of study, patients are follow-up for 3 months.

ELIGIBILITY:
Inclusion Criteria:

* Aged 18 and over
* Sufficiently fluent in English
* On active treatment receiving systemic therapy (e.g., chemotherapy, immunotherapy, hormonal therapy, etc.) or radiotherapy
* Patients with diagnosis of a genitourinary (GU) cancer (e.g., prostate, kidney, and bladder cancer) who have grade 1 or 2 fatigue based on physician assessment at the time of study entry
* Clinician assessed prognosis of greater than or equal to six months
* Willing and independently able to provide consent
* Receive a pre-screen FACIT-Fatigue score of less than or equal to 30

Exclusion Criteria:

* Severe sleep disorders (e.g. narcolepsy)
* Eye Diseases which limit the ability of light to be processed (e.g. untreated cataracts, severe glaucoma, macular degeneration, blindness, pupil dilation problems or other retinal disorder)
* Severe psychological impairment (e.g., bipolar disorder or manic episodes)
* Current employment in night shift work
* Previous use of light therapy to alleviate fatigue or depressive symptoms
* Secondary cancer diagnosis within the past 5 years
* Plans to travel across meridians during treatment
* Pregnancy
* Currently recovering from previous eye surgery within the past 6 months that causes eye irritation
* Sensitivity to light, epilepsy, or a history of seizures

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 224 (Estimated)
Dates: Start 2022-11-29 (Actual); Primary Completion 2027-05-25 (Estimated); Study Completion 2027-05-25 (Estimated)

PRIMARY OUTCOMES:
Functional Assessment of Cancer Therapy - (FACIT) | At baseline
  The effects of light therapy and occupational therapy (OT) on FACIT will be evaluated by comparing light therapy to no-light therapy and comparing occupational therapy to no-occupational therapy. Analysis of variance test will be used for the factorial comparisons, with a two-sided statistical significance level (alpha = 0.05). The interaction between occupational therapy and light therapy will be explored (to understand whether the effect of light therapy [if any] on FACIT would change with occupational therapy and vice versa). The Functional Assessment of Chronic Illness Therapy (FACIT- fatigue scale) is a 13-item patient-reported measure of fatigue. Items are scored on a 0 - 4 response scale with anchors ranging from "Not at all" to "Very much so". To score the FACIT-fatigue, all items are summed to create a single fatigue score with a range from 0 to 52. The higher the score, the better the Quality of Life (QoL).
Functional Assessment of Cancer Therapy - (FACIT) | 6 weeks after baseline
  The effects of light therapy and occupational therapy (OT) on FACIT will be evaluated by comparing light therapy to no-light therapy and comparing occupational therapy to no-occupational therapy. Analysis of variance test will be used for the factorial comparisons, with a two-sided statistical significance level (alpha = 0.05). The interaction between occupational therapy and light therapy will be explored (to understand whether the effect of light therapy [if any] on FACIT would change with occupational therapy and vice versa). The Functional Assessment of Chronic Illness Therapy (FACIT- fatigue scale) is a 13-item patient-reported measure of fatigue. Items are scored on a 0 - 4 response scale with anchors ranging from "Not at all" to "Very much so". To score the FACIT-fatigue, all items are summed to create a single fatigue score with a range from 0 to 52. The higher the score, the better the Quality of Life (QoL).
Functional Assessment of Cancer Therapy - (FACIT) | 3 months after baseline
  The effects of light therapy and occupational therapy (OT) on FACIT will be evaluated by comparing light therapy to no-light therapy and comparing occupational therapy to no-occupational therapy. Analysis of variance test will be used for the factorial comparisons, with a two-sided statistical significance level (alpha = 0.05). The interaction between occupational therapy and light therapy will be explored (to understand whether the effect of light therapy [if any] on FACIT would change with occupational therapy and vice versa). The Functional Assessment of Chronic Illness Therapy (FACIT- fatigue scale) is a 13-item patient-reported measure of fatigue. Items are scored on a 0 - 4 response scale with anchors ranging from "Not at all" to "Very much so". To score the FACIT-fatigue, all items are summed to create a single fatigue score with a range from 0 to 52. The higher the score, the better the Quality of Life (QoL).

SECONDARY OUTCOMES:
Longitudinal change in FACIT-Fatigue scores | Baseline
  Will evaluate whether the longitudinal change in FACIT-Fatigue scores, is significantly different between the intervention groups, including the control group. The Functional Assessment of Chronic Illness Therapy (FACIT- fatigue scale) is a 13-item patient-reported measure of fatigue. Items are scored on a 0 - 4 response scale with anchors ranging from "Not at all" to "Very much so". To score the FACIT-fatigue, all items are summed to create a single fatigue score with a range from 0 to 52. The higher the score, the better the QoL.
Longitudinal change in FACIT-Fatigue scores | 6 weeks after baseline
  Will evaluate whether the longitudinal change in FACIT-Fatigue scores, is significantly different between the intervention groups, including the control group. The Functional Assessment of Chronic Illness Therapy (FACIT- fatigue scale) is a 13-item patient-reported measure of fatigue. Items are scored on a 0 - 4 response scale with anchors ranging from "Not at all" to "Very much so". To score the FACIT-fatigue, all items are summed to create a single fatigue score with a range from 0 to 52. The higher the score, the better the QoL.
Longitudinal change in FACIT-Fatigue scores | 3 months after baseline
  Will evaluate whether the longitudinal change in FACIT-Fatigue scores, is significantly different between the intervention groups, including the control group. The Functional Assessment of Chronic Illness Therapy (FACIT- fatigue scale) is a 13-item patient-reported measure of fatigue. Items are scored on a 0 - 4 response scale with anchors ranging from "Not at all" to "Very much so". To score the FACIT-fatigue, all items are summed to create a single fatigue score with a range from 0 to 52. The higher the score, the better the QoL.
Self-reported occupational performance - Baseline | Baseline
  Will determine if an OT-based intervention can improve self-reported occupational performance from preassessment to immediately after time point 2 (session 6) This outcome measure is Canadian Occupational Performance Measure (COPM). Its administration involves four steps: (a) the patient is asked to identify occupations that are difficult for him or her in self-care, productivity and leisure; (b) the importance of these problem occupations is rated on a scale of 1-10 in terms of importance (1 = least important, 10 = most important); (c) patients' perceptions of performance and satisfaction with their five most important problems are rated on two separate 10-point scales (performance 1 = not able to do it, 10 = able to do it extremely well; satisfaction 1 = not satisfied at all, 10 = extremely satisfied) and finally (d) at reassessment both the performance and satisfaction ratings are repeated (and the change between assessment and reassessment is evaluated).
Self-reported occupational performance - session 6 | 6 weeks after baseline
  Will determine if an OT-based intervention can improve self-reported occupational performance from preassessment to immediately after time point 2 (session 6) This outcome measure is Canadian Occupational Performance Measure (COPM). Its administration involves four steps: (a) the patient is asked to identify occupations that are difficult for him or her in self-care, productivity and leisure; (b) the importance of these problem occupations is rated on a scale of 1-10 in terms of importance (1 = least important, 10 = most important); (c) patients' perceptions of performance and satisfaction with their five most important problems are rated on two separate 10-point scales (performance 1 = not able to do it, 10 = able to do it extremely well; satisfaction 1 = not satisfied at all, 10 = extremely satisfied) and finally (d) at reassessment both the performance and satisfaction ratings are repeated (and the change between assessment and reassessment is evaluated).

CONTACTS AND LOCATIONS:
Overall Officials: William Dale, Principal Investigator — City of Hope Medical Center
Locations (1):
- City of Hope Medical Center, Duarte, California, United States